CLINICAL TRIAL: NCT03326713
Title: Comparative Effectiveness of Interventions to Increase Guideline-based Genetic Counseling in Ethnically and Geographically Diverse Cancer Survivors
Brief Title: Genetic Risk Assessment for Cancer Education and Empowerment (GRACE) Project
Acronym: GRACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Colorado Department of Public Health and Environment (Other Government); University of New Mexico (Other)
Responsible Party: Principal Investigator, Anita Y. Kinney, PhD, RN, Study Principal Investigator; Associate Director for Cancer Health Equity, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro2018001350
Record Dates: First submitted 2017-10-17; First posted 2017-10-31 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Ovarian Cancer
Keywords: Genetic Testing; Prevention
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: 3-arm Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Randomization will be single blinded. Research team members who are assessing the outcomes will be blinded to study arm assignment. Research staff who are conducting follow-up interviews will be blinded to group assignment as much as possible. At the beginning of the follow-up interviews, the interviewer will request that the participant does not reveal the study arm they were assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telephone Counseling & Navigation (TCN) (Experimental): Telephone Counseling
  Interventions: Behavioral: Telephone Counseling & Navigation (TCN)
- Mailed Targeted Print (TP) (Active Comparator): Mailed Targeted Print
  Interventions: Behavioral: Mailed Targeted Print (TP)
- Usual Care (UC) (Other): Control
  Interventions: Other: Usual Care (UC)

INTERVENTIONS:
Behavioral: Telephone Counseling & Navigation (TCN) — A health coach will conduct a 30-45 minute telephone counseling session with participants. Prior to the telephone session, participants will receive the same brochure that the TP arm receives. After the phone call, participants will receive a tailored follow-up letter which will include images tailored to the individual's age, self-identified ethnicity, and family composition.
  Arms: Telephone Counseling & Navigation (TCN)
Behavioral: Mailed Targeted Print (TP) — Participants will be mailed an educational brochure within two weeks of completing the baseline survey that addresses important evidence-based theoretical targets: CGRA guideline (knowledge), threat appraisal (to validate or raise risk perceptions, HBOC seriousness), response efficacy (benefits and expectations about CGRA), self-efficacy messages (CGRA resources, insurance reimbursement, and assistance for those with financial challenges) and possible actions to take (make an appointment and discuss with provider). Both the targeted print and tailored intervention materials were developed using formative community engaged research methods.
  Arms: Mailed Targeted Print (TP)
Other: Usual Care (UC) — A usual care arm is included to assess CGRA uptake in the absence of intervention as well as priming from the surveys for the primary outcome analysis.
  Arms: Usual Care (UC)

SUMMARY:
GRACE is a randomized 3-arm trial to determine the comparative effectiveness of two remote cancer communication interventions: 1) a targeted generic print (TP) or 2) a tailored telephone-based counseling and navigation intervention (TCN). Post-award, the target sample size was revised to (n=642) with NIH permission.

DETAILED DESCRIPTION:
There is increasing evidence that activated and engaged patients who are equipped with necessary skills and information are more likely to follow through with recommended care and have better health outcomes at reduced costs. Identification of individuals at increased risk of hereditary breast and ovarian cancer (HBOC) is crucial for cancer survivors and their families to benefit from biomedical advances in cancer prevention, early detection, treatment and survivorship. The primary purpose of this study is to assess the feasibility and acceptability of two remote interventions aimed at promoting cancer genetic risk assessment (CGRA) for HBOC. The randomized controlled trial will have 3 arms: usual care (UC) vs. targeted generic print (TP) vs. tailored telephone counseling and navigation intervention (TCN).

ELIGIBILITY:
Inclusion Criteria:

Breast Cancer

* Hispanic or non-Hispanic
* Female
* 21 years of age or older
* English-speaking
* Breast cancer history

  * breast cancer at the age of 50 or younger OR
  * triple-negative breast cancer OR
  * two or more primary breast cancers

Ovarian Cancer

* Hispanic or non-Hispanic
* Female
* 21 years of age or older
* English-speaking
* History of ovarian, fallopian, or peritoneal cancer diagnosed at any age

Exclusion Criteria:

Have had prior genetic counseling or testing for hereditary breast and/or ovarian cancer

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita Y Kinney, PhD, RN, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] An J, McDougall J, Lin Y, Lu SE, Walters ST, Heidt E, Stroup A, Paddock L, Grumet S, Toppmeyer D, Kinney AY. Randomized trial promoting cancer genetic risk assessment when genetic counseling cost removed: 1-year follow-up. JNCI Cancer Spectr. 2024 Feb 29;8(2):pkae018. doi: 10.1093/jncics/pkae018. PMID 38490263
- [Derived] Kinney AY, Walters ST, Lin Y, Lu SE, Kim A, Ani J, Heidt E, Le Compte CJG, O'Malley D, Stroup A, Paddock LE, Grumet S, Boyce TW, Toppmeyer DL, McDougall JA. Improving Uptake of Cancer Genetic Risk Assessment in a Remote Tailored Risk Communication and Navigation Intervention: Large Effect Size but Room to Grow. J Clin Oncol. 2023 May 20;41(15):2767-2778. doi: 10.1200/JCO.22.00751. Epub 2023 Feb 14. PMID 36787512
- [Derived] Le Compte CG, Lu SE, Ani J, McDougall J, Walters ST, Toppmeyer D, Boyce TW, Stroup A, Paddock L, Grumet S, Lin Y, Heidt E, Kinney AY. Understanding cancer genetic risk assessment motivations in a remote tailored risk communication and navigation intervention randomized controlled trial. Health Psychol Behav Med. 2022 Dec 9;10(1):1190-1215. doi: 10.1080/21642850.2022.2150623. eCollection 2022. PMID 36518606
- [Derived] Kinney AY, Blair CK, Guest DD, Ani JK, Harding EM, Amorim F, Boyce T, Rodman J, Ford CG, Schwartz M, Rosenberg L, Foran O, Gardner J, Lin Y, Arap W, Irwin MR. Biobehavioral effects of Tai Chi Qigong in men with prostate cancer: Study design of a three-arm randomized clinical trial. Contemp Clin Trials Commun. 2019 Aug 21;16:100431. doi: 10.1016/j.conctc.2019.100431. eCollection 2019 Dec. PMID 31650067
- [Derived] Kinney AY, Howell R, Ruckman R, McDougall JA, Boyce TW, Vicuna B, Lee JH, Guest DD, Rycroft R, Valverde PA, Gallegos KM, Meisner A, Wiggins CL, Stroup A, Paddock LE, Walters ST. Promoting guideline-based cancer genetic risk assessment for hereditary breast and ovarian cancer in ethnically and geographically diverse cancer survivors: Rationale and design of a 3-arm randomized controlled trial. Contemp Clin Trials. 2018 Oct;73:123-135. doi: 10.1016/j.cct.2018.09.005. Epub 2018 Sep 18. PMID 30236776

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 3 statewide cancer registries in New Jersey, Colorado, and New Mexico between November 2017 and July 2020.
Pre-assignment Details: 668 met inclusion criteria, were enrolled and randomized, and 658 received their assigned intervention.
Groups:
- Usual Care (UC): Included to assess CGRA uptake without intervention and to provide context for the primary outcome analysis.
- Tailored Print (TP): Mailed Targeted Print:
  Participants received an educational brochure within two weeks of completing the baseline survey. This brochure addressed key evidence-based targets: CGRA guidelines, threat appraisal, response efficacy, self-efficacy messages, and actionable steps (e.g., making an appointment). The materials were developed through community-engaged research methods.
- Tailored Counseling & Navigation (TCN): Telephone Counseling:
  A health coach conducted a 30-45 minute telephone counseling session with participants. Before the call, they received the same brochure as the TP arm. After the session, participants received a personalized follow-up letter featuring images tailored to their age, self-identified ethnicity, and family composition.
Period: Overall Study
Arm/Group | Usual Care (UC) | Tailored Print (TP) | Tailored Counseling & Navigation (TCN)
Started | 223 | 225 | 220
Received Intervention | 223 | 224 | 211
Completed | 189 | 190 | 168
Not Completed | 34 | 35 | 52
Not completed — Death | 2 | 1 | 0
Not completed — Lost to Follow-up | 20 | 21 | 33
Not completed — Withdrawal by Subject | 1 | 2 | 11
Not completed — Found Ineligible | 11 | 11 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All randomized participants who remained eligible.
Groups:
- Mailed Targeted Print (TP): Mailed Targeted Print:
  Participants receive an educational brochure within two weeks of completing the baseline survey. This brochure addresses key evidence-based targets: CGRA guidelines, threat appraisal, response efficacy, self-efficacy messages, and actionable steps (e.g., making an appointment). The materials were developed through community-engaged research methods.
- Tailored Counseling & Navigation (TCN): Telephone Counseling:
  A health coach will conduct a 30-45 minute telephone counseling session with participants. Before the call, they will receive the same brochure as the TP arm. After the session, participants will receive a personalized follow-up letter featuring images tailored to their age, self-identified ethnicity, and family composition.
- Total: Total of all reporting groups
Arm/Group | Usual Care (UC) | Mailed Targeted Print (TP) | Tailored Counseling & Navigation (TCN) | Total
Number analyzed (Participants) | 212 | 214 | 212 | 638
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (10.0) | 61.0 (10.1) | 61.2 (10.7) | 61.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 214 | 212 | 638
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 46 | 58 | 159
  Not Hispanic or Latino | 152 | 165 | 150 | 467
  Unknown or Not Reported | 5 | 3 | 4 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 3 | 7
  Asian | 9 | 7 | 11 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 18 | 14 | 39
  White | 160 | 153 | 148 | 461
  More than one race | 5 | 15 | 5 | 25
  Unknown or Not Reported | 29 | 19 | 31 | 79
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Mid-Atlantic, United States | 62 | 59 | 63 | 184
  United States: West, United States | 41 | 56 | 37 | 134
  United States: Southwest, United States | 109 | 99 | 112 | 320
Years Since Diagnosis [Mean (Standard Deviation); unit: years] — Number of years elapsed since a participant was diagnosed with cancer.
  years | 11.3 (7.7) | 10.9 (7.6) | 11.3 (7.7) | 11.2 (7.7)
Annual Household Income [Count of Participants; unit: Participants] — Total income earned by all members of a household within a year.
  Participants
    <$30,000 | 51 | 43 | 46 | 140
    $30,000-$49,999 | 35 | 35 | 31 | 101
    $50,000-$69,999 | 29 | 28 | 28 | 85
    $70,000 or more | 73 | 84 | 83 | 240
    Missing | 24 | 24 | 24 | 72
Education Level [Count of Participants; unit: Participants] — Participant highest completed level of education.
  Participants
    Less than high school/High school grad/GED | 43 | 40 | 32 | 115
    Some college, associate degree, or vocational school | 80 | 67 | 80 | 227
    Bachelor's degree or higher | 88 | 105 | 97 | 290
    Missing | 1 | 2 | 3 | 6
Health Insurance [Count of Participants; unit: Participants] — Whether a participant has health insurance coverage at the time of data collection.
  Participants
    Does not have health insurance | 15 | 7 | 12 | 34
    Has health insurance | 197 | 207 | 198 | 602
    Missing | 0 | 0 | 2 | 2
Cancer Site [Count of Participants; unit: Participants] — Specific location or organ in the body where participant cancer originates.
  Participants
    Ovarian | 36 | 32 | 26 | 94
    Breast | 176 | 182 | 186 | 544
Language Preference [Count of Participants; unit: Participants] — Participant preferred language for communication.
  Participants
    English | 196 | 211 | 204 | 611
    Spanish | 16 | 3 | 8 | 27
Health Literacy Level [Count of Participants; unit: Participants] — Assessed with a validated measure used to screen for people with inadequate health literacy. Response options are scored on a Likert scale of 0-4. Items are summed for a maximum health literacy score of 12.
  Participants
    Adequate (<9) | 208 | 208 | 208 | 624
    Marginal/Inadequate (greater than or equal to 9) | 4 | 5 | 4 | 13
    Missing | 0 | 1 | 0 | 1
Family History of Cancer [Count of Participants; unit: Participants] — Number of first-degree relatives (FDR) and second-degree relatives (SDR) with breast or ovarian cancer
  Participants
    0 FDR and 0 SDR | 131 | 140 | 135 | 406
    1 FDR or 1 SDR | 49 | 40 | 42 | 131
    2 or more FDR/SDR | 32 | 34 | 35 | 101
Marital Satus [Count of Participants; unit: Participants] — Participant current marital status at time of data collection.
  Participants
    Single/Divorced/Separated/Widowed | 76 | 88 | 85 | 249
    Married/Domestic partnership | 136 | 125 | 127 | 388
    Missing | 0 | 1 | 0 | 1
Has a Personal Healthcare Provider [Count of Participants; unit: Participants] — Whether participant has a designated personal healthcare provider, such as a primary care physician.
  Participants
    No does not have a personal healthcare provider | 9 | 8 | 9 | 26
    Yes has a personal healthcare provider | 203 | 206 | 203 | 612
Informed of Increased HBOC Risk by Healthcare Provider [Count of Participants; unit: Participants] — Whether participant has been informed by a healthcare provider about their increased risk for hereditary breast and ovarian cancer (HBOC).
  Participants
    No | 133 | 130 | 122 | 385
    Yes | 79 | 83 | 90 | 252
    Missing | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Medically Verified Cancer Genetic Risk Assessment Uptake at 6 Months
Description: Participants reported whether they had sought cancer CGRA (i.e. genetic counseling and/or testing) in surveys at the 6-month follow-up. Participants who reported receiving a CGRA were asked to provide written consent allowing research staff to obtain document of receipt of the genetic services.
Time Frame: 6 months following the interventions for TP and TCN, and 6 months following the baseline survey for the UC arm.
Population: Eligible participants analyzed at 6 months.
Measure: Count of Participants; unit: Participants
Groups:
- Tailored Counseling and Navigation (TCN): Telephone Counseling:
  A health coach conducted a 30-45 minute telephone counseling session with participants. Before the call, they received the same brochure as the TP arm. After the session, participants received a personalized follow-up letter featuring images tailored to their age, self-identified ethnicity, and family composition.
Arm/Group | Usual Care (UC) | Tailored Print (TP) | Tailored Counseling and Navigation (TCN)
Number analyzed (Participants) | 213 | 216 | 212
Participants | 5 | 6 | 32
Statistical Analysis 1: Comparison: Tailored Print (TP) vs Tailored Counseling and Navigation (TCN); Logistic Regression Model Results for Intervention Effects on CGRA Within 6 Months (TP vs TCN); Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 6.2, 95% CI 2-sided [2.5 to 15.2]
Statistical Analysis 2: Comparison: Usual Care (UC) vs Tailored Counseling and Navigation (TCN); Logistic Regression Model Results for Intervention Effects on CGRA Within 6 Months (UC vs TCN); Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 7.4, 95% CI 2-sided [2.8 to 19.4]
Statistical Analysis 3: Comparison: Usual Care (UC) vs Tailored Print (TP); Logistic Regression Model Results for Intervention Effects on CGRA Within 6 Months (UC vs TP); Test type: Superiority; p = 1.2, Regression, Logistic; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.4 to 4.0]

2. Secondary Outcome: Medically Verified Cancer Genetic Risk Assessment Uptake at 12 Months
Description: Participants reported whether they had sought cancer CGRA (i.e. genetic counseling and/or testing) in surveys at the 12-month follow-up. Participants who reported receiving a CGRA were asked to provide written consent, allowing research staff to obtain documents of receipt of the genetic services.
Time Frame: 12 months following the interventions for TP and TCN, and 12 months following the baseline survey for the UC arm.
Population: Eligible participants analyzed at 12-months.
Measure: Count of Participants; unit: Participants
Groups:
- Tailored Print (TP): Mailed Targeted Print:
  Participants receive an educational brochure within two weeks of completing the baseline survey. This brochure addresses key evidence-based targets: CGRA guidelines, threat appraisal, response efficacy, self-efficacy messages, and actionable steps (e.g., making an appointment). The materials were developed through community-engaged research methods.
Arm/Group | Usual Care (UC) | Tailored Print (TP) | Tailored Counseling & Navigation (TCN)
Number analyzed (Participants) | 212 | 214 | 212
Participants | 23 | 21 | 45

3. Secondary Outcome: Decisional Conflict for CGRA: SURE Scale
Description: Questionnaire: Decisional conflict associated with the CGRA decision will be measured separately with 4 items using the SURE Scale (Sure of myself; Understand information; Risk-benefit ratio; Encouragement). Range from 0-4, with 0 indicating high decisional conflict.
Time Frame: 1 month following the interventions for TP and TCN, and 1 months following the baseline survey for the UC arm.
Population: Eligible participants analyzed at 1 month.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Tailored Print (TP) | Tailored Counseling & Navigation (TCN)
Number analyzed (Participants) | 213 | 216 | 212
score on a scale | 2.44 (2.11) | 2.55 (1.79) | 3.33 (1.16)

4. Secondary Outcome: Cancer Genetic Risk Assessment Intention
Description: Questionnaire: One item will measure future intention to get a cancer genetic risk assessment within the next 6 weeks. Responses for this item ranged from 1 (not at all) to 5 (extremely likely).
Time Frame: 1 month following the interventions for TP and TCN, and 1 months following the baseline survey for the UC arm.
Population: Eligible participants analyzed at 1 month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care (UC) | Tailored Print (TP) | Tailored Counseling & Navigation (TCN)
Number analyzed (Participants) | 213 | 216 | 212
units on a scale | 2.69 (1.27) | 2.78 (1.29) | 3.44 (1.46)

ADVERSE EVENTS:
Time Frame: Time of enrollment through study completion, an average of 13 months.
Description: The study is of minimal risk to participants. Adverse events were self-reported through surveys and during communications with research personnel.
Arm/Group | Usual Care (UC) | Tailored Print (TP) | Tailored Counseling & Navigation (TCN)
All-Cause Mortality (participants affected / at risk) | 2/223 | 1/225 | 0/220
Serious Adverse Events (participants affected / at risk) | 0/223 | 0/225 | 0/220
Other Adverse Events (participants affected / at risk) | 0/223 | 0/225 | 0/220

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-11-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT03326713/Prot_001.pdf
  • Statistical Analysis Plan (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/13/NCT03326713/SAP_002.pdf
  • Informed Consent Form (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT03326713/ICF_000.pdf